CLINICAL TRIAL: NCT03650621
Title: Magnetic Non-Invasive Acupuncture For Infant Comfort A Pilot Study in Preterm Infants Requiring Eye-exam for Retinopathy of Prematurity
Brief Title: Acupuncture for Preterm Infants Requiring Eye-exam
Acronym: MAGNIFIC-ROP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00080714
Record Dates: First submitted 2018-06-26; First posted 2018-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-07

CONDITIONS: Retinopathy of Prematurity; Pain; Acupuncture; Premature Infant
MeSH Terms: conditions — Retinopathy of Prematurity; Pain; Premature Birth

STUDY DESIGN:
Intervention Model Description: this is a 2-arm parallel design randomized controlled trial with 3 sites recruiting infants
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: patients are preterm infants and therefore mask, health care providers will be masked as well as outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Magnetic acupuncture (Experimental): Infants randomized to the intervention arm will have 5 magnetic stickers placed on both ears approximately 1 hour before the eye-exam and will stay in place for approximately 1 hour after the eye-exam.
  Total duration of study 2.5-3 hours
  Interventions: Device: Magnetic acupuncture
- Control - Placebo control (Placebo Comparator): In this arm the infants will have 5 stickers (magnets removed) placed on their ear approximately 1 hour before the eye-exam and will stay in place for approximately 1 hour after the eye-exam.
  Total duration of study 2.5-3 hours
  Interventions: Device: stickers (magnets removed)

INTERVENTIONS:
Device: Magnetic acupuncture — 5 magnetic acupuncture stickers will be placed on the infants ear
  Arms: Intervention - Magnetic acupuncture
Device: stickers (magnets removed) — in this group 5 stickers (magnets removed) will be placed on the infants ear
  Arms: Control - Placebo control

SUMMARY:
The purpose is to investigate whether non-invasive acupuncture - NIA (i.e. acupuncture without needles) will help reduce pain for babies in the Neonatal Intensive Care Unit (NICU) during their routine weekly eye-exam for Retinopathy of prematurity. Retinopathy of prematurity (ROP) is an eye disease most commonly affecting premature babies born weighing less than 1250 grams. Retinopathy of prematurity occurs because these premature babies require oxygen because of their immature lungs. The oxygen then stimulates the growth of blood vessels in the retina, causing the retina to be detached from the eye, which causes vision impairment.

To examine if the vessels grow at the back of the eye, an eye-doctor visits bi-weekly once the baby is 32 weeks corrected age to assess if the blood vessels change. If there is a lot of growth, the eye-doctor would use a laser to treat the eye to prevent further growth.

During the bi-weekly eye-exam, the premature infant receives sucrose (a type of sugar) for pain management. The investigator will assess pain a premature babies experience during this exam and found that there are extremely high scores of pain despite sucrose and the investigator believe this pain and stress caused by these procedures could be reduced by adding:

Magnetic Acupuncture

Also, untreated pain causes stress (lower oxygen levels, higher heart rates), discomfort and poorer long term outcomes.

Finding the best treatment and prevention for the pain caused by procedures in the NICU is therefore extremely important for any baby.

DETAILED DESCRIPTION:
Background: Infants in neonatal intensive care units (NICU) may experience as many as 14 painful and stressful procedures every day. Even common and seemingly innocuous procedures like routine eye exams can cause relatively severe pain that is only marginally alleviated by powerful analgesics like morphine. Infants subject to severe and repeated episodes of pain are at risk of immediate and long-term sequelae, including intraventricular hemorrhage, impaired neurodevelopment, poor postnatal growth, cognitive and motor dysfunction and emotional dysregulation. Pharmacological analgesia is often used in the NICU to either prevent or alleviate procedural pain but none are completely effective and almost all have potentially detrimental side-effects. Non-pharmacological measures (e.g., kangaroo care and breastfeeding) are also used but these methods may not be feasible in very sick infants or if pain is extremely severe. Methods to provide safe and effective analgesia for babies in the NICU are therefore needed. Acupuncture has been used for thousands of years to prevent and treat pain and various health conditions. There are many forms of acupuncture, including needling, electrical currents, laser, and pressure, all of which aim to modulate activity of key nociceptive structures, neurotransmitter secretions and parasympathetic function. The investigator have reported about the safety and efficacy of auricular magnetic acupuncture (MA) in the NICU environment during heel pricks or neonatal withdrawal. One of the most common and painful procedure preterm infants experience during their NICU stay is their weekly eye-exam to assess for Retinopathy of Prematurity. Currently, during the eye exam infants receive sucrose for analgesia, which has very limited effects on pain release. The investigator propose to examine if using auricular MA will reduce pain during their eye-exam.

Research question: Does auricular MA decrease pain in preterm infants compared to placebo with control.

Aim: To determine if auricular MA will reduce pain compared to placebo with control in preterm infants during their eye exam.

Hypothesis: The investigator hypotheses that auricular MA will reduce pain compared to placebo with control in preterm infants during their eye exam.

Methods: Infants who will require their routine eye exam (beginning at 32 weeks corrected age) will be randomized to either auricular MA or auricular placebo/sucrose after parental informed consent. Five auricular MA or placebo stickers will be placed on acupuncture sites on both ears for 1 hour prior to the eye-exam by a non-blinded investigator. Pain responses will be assessed with the Premature Infant Pain Profile (PIPP) by blinded clinicians before, during and after each eye-exam. The study will be conducted in the NICU at the Royal Alexandra Hospital as a single-blinded randomized, placebo controlled study to investigate the safety and feasibility of using magnetic stickers in the NICU environment. The randomization sequence will be pre-specified, computer generated into block sizes of 2-4. Allocations will be concealed in sequential opaque envelopes stored in a secure location. A single unblinded investigator will complete randomization, administer the intervention, but will not be involved in data collection. Infants will be randomized to receive either MA or placebo stickers that are to be applied bilaterally to the 5 auricular acupuncture points as per the Battlefield Acupuncture (BFA) protocol at least 1 hour prior to the eye-exam by the unblinded investigator. Placebos will be constructed by removing the magnet ball from pre commercially-available MA plasters (Sakamura, Helio Acupuncture, Japan). The magnet site on placebo and magnetic stickers will then be concealed with a thick application of white, opaque correction fluid. Stickers will be removed 1 hour after the eye-exam. Sucrose for pain management can be given as per NICU policy. The ROP eye exams are performed by a dedicated group of five physicians therefore consistency will be maintained. Primary outcome: Infant's response to the pain during the eye-exam, measured by the PIPP score, a validated, quantitative pain assessment tool for use in premature infants.

Expected outcomes: The proposed study aims to examine if auricular MA compared to placebo will decrease pain in premature infants. If validated, the results of the study could be translated into NICUs around the world and might benefit a large number of babies each year.

ELIGIBILITY:
Inclusion Criteria:

* Infants weighing less than 1250g at birth admitted into the NICU at the Royal Alexandra Hospital will require routine,regularly scheduled ROP eye-exams beginning at 32 weeks corrected age. We will not enroll any infant who meets any exclusion criteria.

Exclusion Criteria:

1. Chronic pain stimuli (e.g. infants who have had recent surgery)
2. Neurological problems that could impair pain perception (e.g. diagnosis of intraventricular hemorrhages Grade III or greater)
3. Cardiorespiratory problems that could impair oxygenation (e.g. any infant who is intubated and requiring mechanical ventilation)

Ages: 29 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in Premature Infant Pain Profile (PIPP) scores | Comparison of baseline (= 1 hour before eye-exam) and after eye-exam (1 hour after)
  Mean pain scores on the Premature Infant Pain Profile (PIPP) scores

SECONDARY OUTCOMES:
Heart rate changes | changes in heart rate in beats per minute 1 hour before and 1 hour after eye-exam
  During eye-exam - which will take 5min (comparison between baseline before eye-exam and mean value during eye-exam)
Changes in oxygen saturation | changes in oxygen saturation in % 1 hour before and 1 hour after eye-exam
  During eye-exam - which will take 5min (comparison between baseline before eye-exam and mean value during eye-exam)
changes in cerebral oxygenation | changes in cerebral oxygenation % 1 hour before and 1 hour after eye-exam
  During eye-exam - which will take 5min (comparison between baseline before eye-exam and mean value during eye-exam)

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, MD, PhD, Principal Investigator — University of Alberta
Locations (3):
- University of Sydney, Sydney, New South Wales, Australia
- Royal Alexandra Hospital, Edmonton, Alberta, Canada
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: once study has been completed
Access Criteria: email to PI

REFERENCES:
- [Derived] Gan KML, Oei JL, Quah-Smith I, Kamar AA, Lordudass AAD, Liem KD, Lindrea KB, Daly M, Gaunker N, Mangat AK, Yaskina M, Schmolzer GM. Magnetic Non-invasive Auricular Acupuncture During Eye-Exam for Retinopathy of Prematurity in Preterm Infants: A Multicentre Randomized Controlled Trial. Front Pediatr. 2020 Dec 23;8:615008. doi: 10.3389/fped.2020.615008. eCollection 2020. PMID 33425820